CLINICAL TRIAL: NCT01080729
Title: A Prospective, Observational and Multicentric Study to Compare the Dose of GONAL-fTM FbM Prescribed by the Doctor With the Recommendation of the Dose Calculator Consort and to Evaluate the Ease of Use of Pre-filled Pen of GONAL-fTM FbM Pen
Brief Title: An Observational Study to Compare the Dose of Gonal-fTM FbM Prescribed by the Doctor With the Recommendation of the Dose Calculator Consort and to Evaluate the Ease of Use of Pre-filled Pen of Gonal-fTM FbM Pen
Status: Terminated | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck N.V.-S.A., Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: 700623-508
Record Dates: First submitted 2010-03-03; First posted 2010-03-04 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2011-10

CONDITIONS: Multifollicular Stimulation
Keywords: Ovulation induction; Ovarian Hyperstimulation Syndrome; Multifollicular stimulation; Pregnancy; Sperm injections, intracytoplasmic; Fertility
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Glycoprotein Hormones, alpha Subunit; follitropin alfa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Serum
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Recombinant-follicle stimulating hormone (r-FSH) — The dosage and administration of r-FSH will be in accordance with the PFS and current clinical practice in the centers (300 IU/0.5 ml [22 micrograms/0.5 ml]; 450 IU/0.75 ml [33 micrograms/0.75 ml]; or 900 IU/1.5 ml [66 micrograms/1.5 ml].
  The dosage and administration of recombinant-hCG (r-hCG; 250 micrograms/0.5 ml), injectable solution in a pre-filled syringe will also be in accordance with the PFS and current clinical practice in the centers (only if the doctor decides to start treatment with r-hCG).
  Other Names: GONAL-f™

SUMMARY:
This is a prospective, observational and multicentric study to compare the Gonal-f FbM (filled by mass) dose prescribed by the doctor with the Gonal-f FbM dose determined by the CONSORT (Consistency in r-FSH Starting doses for individualized treatment) calculator.

DETAILED DESCRIPTION:
The ovarian stimulation with the follicle-stimulating hormone (FSH) is the main element for the success of medically assisted procreation (MAP) technique. The possibility of predicting a poor ovarian response would thus enable the doctor to proactively define the treatment cycle and subject expectations. However, it is difficult to select the right dose of recombinant-human FSH (r-hFSH) to reach the "acceptable" number of oocytes. A series of reports, in which investigators identified different variables associated with ovarian response, appeared in the literature so as to develop a more structured approach with the aim of determining the initial Gonal-f dose in an MAP cycle.

After having reviewed the literature, following predictive factors present a strong correlation with the ovarian response:

* Initial serum FSH during the premature follicle phase (day 2-4 of the cycle),
* Body mass index (BMI; in kg/m2),
* Age,
* Initial number of antral follicles (day 2-4 of the cycle) determined in the ultrasound scan.

The relative importance of each of these factors was judged on the basis of a statistical model analysis and an r-hFSH dose (Gonal-f in international units [IU]) was attributed to each factor with a view of creating guidelines and determining the optimal FSH dose (using CONSORT dose calculator) to be used on the basis of the initial predictive characteristics/variables specific to the subject.

The purpose of this study is to compare the Gonal-f FbM dose prescribed by the doctor with the Gonal-f FbM dose determined by the CONSORT calculator.

A short questionnaire will be used to evaluate the ease of using the pre-filled Gonal-f (FbM) pen. The dosage and administration of Gonal-f shall be in accordance with the Product Features Summary (PFS) and current clinical practice in the centers.

OBJECTIVES

Primary objective:

* To study whether the Gonal-f FbM dose prescribed by the doctor is different from the dose recommended by the CONSORT dose calculator

Secondary objectives:

* To evaluate the ease of using the new generation Gonal-f pen for subjects
* To compare the Gonal-f dose finally used with the dose used during the previous treatment cycles (if this data is available)
* To put a figure to the total duration of the treatment, total quantity of gonadotropins taken and the number of clinical pregnancies
* In case of use of the CONSORT calculator: to estimate cancellations due to poor response This observational study will be conducted in 8 fertility centers in Belgium and Luxembourg as per the current clinical practice conditions in force at each center. Each center will recruit approximately 30 subjects to reach a total of approximately 250 subjects. The maximum number of treatment cycles to be evaluated in this project will be 600 over a period of approximately 6 months.

The CONSORT dose calculator is made available to all the participating centers via a secure web site. Each investigator will receive a user identification and password to access the system. The investigator will then introduce the 4 individual variables of the subject (basal FSH, BMI, age and number of antral follicles [follicles ≥2mm - <11mm]) in the CONSORT calculator, which will determine an individualized dose of Gonal-f for this specific subject. If the investigator does not agree with the dose calculated by CONSORT and opts for another dosage, he/she may indicate it directly in the CRF (Case Report Form). In this case, the Gonal-f dose will be based on the investigator's advice in accordance with the clinical practice in force in the center.

Follicle development shall be monitored in accordance with the current clinical practice of the center with diagnostic ultrasound and/or estradiol (E2) dosage until the local criteria for the administration of the human chorionic gonadotropin (hCG) is reached. Human chorionic gonadotropin will be administered in accordance with the current clinical practice of the center to reach final oocyte maturation. The date of administration of the hCG (Ovitrelle) will be indicated in the CRF.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects who started treatment with Gonal-f on the basis of the decision of the investigator and indications and recommendations of the PFS
* Subjects who were at least 35 years old when the Gonal-f dose was administered (i.e. at the time of introducing individual variables of the subject in the CONSORT calculator for determining the dose)
* Subjects with BMI < 30 kg/m2
* Subjects who were in premature follicle phase (day 2-4), basal FSH ≤12 IU/l (measured in the center's laboratory)
* Subjects who were taking a gonadotropin-releasing hormone (GnRH) protocol agonist
* Subjects who consented to participate in the study and inform the investigator about their medical history
* Subjects who signed the written consent form, which stipulated that the subject could dropout of the study at any time without any negative consequences on future medical treatments

Exclusion Criteria:

* Subjects simultaneously participating in an interventional study
* Subjects following concomitant treatment with clomifene citrate
* Subjects presenting one of the contraindications described in the SPC

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female subjects, who are being considered for an IVF/ICSI treatment and a Gonal-f treatment based on the PFS and inclusion and exclusion criteria will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Comparison between the initial Gonal-f FbM dose prescribed by the doctor and the initial Gonal-f FbM dose recommended by the CONSORT calculator | Before and after the treatement for 1 cycle over a period of 6 months

SECONDARY OUTCOMES:
Secondary variables | Before and after the treatement for 1 cycle over a period of 6 months
  Total Gonal-f dose used; subject satisfaction; duration of the treatment; Gonal-f dose used on the last day of stimulation; total dose of gonadotropins used; number of cases of ovarian hyper-stimulation syndrome (OHSS); number of cancelled cycles; number of clinical pregnancies; incidence and seriousness of OHSS

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck N.V.-S.A., Belgium
Locations (1):
- ZNA Middelheim, Antwerp, Lindendreef 1, Belgium